CLINICAL TRIAL: NCT03302234
Title: A Phase 3, Randomized, Double-Blind Study of Pembrolizumab Plus Ipilimumab vs Pembrolizumab Plus Placebo in Previously Untreated, Stage IV, Metastatic Non-small Cell Lung Cancer Subjects Whose Tumors Are PD-L1 Positive (TPS ≥ 50%) (KEYNOTE-598)
Brief Title: Study of Pembrolizumab Given With Ipilimumab or Placebo in Participants With Untreated Metastatic Non-Small Cell Lung Cancer (NSCLC) (MK-3475-598/KEYNOTE-598)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-598; MK-3475-598 (Other: Merck); KEYNOTE-598 (Other: Merck); 2016-004364-20 (EudraCT Number)
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Cytotoxic T-lymphocyte-associated protein 4 (CTLA4); PD1; PD-1; PDL1; PD-L1; CTLA4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — pembrolizumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Ipilimumab (Experimental): Participants receive 200 mg of pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus 1 mg/kg of ipilimumab by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment.
  Interventions: Biological: Pembrolizumab; Biological: Ipilimumab
- Pembrolizumab + Placebo (Active Comparator): Participants receive 200 mg of pembrolizumab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus placebo by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment.
  Interventions: Biological: Pembrolizumab; Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®; MK-3475
Biological: Ipilimumab — Administered as an IV infusion every 6 weeks (Q6W)
  Other Names: YERVOY®
  Arms: Pembrolizumab + Ipilimumab
Other: Placebo — Normal saline solution administered as an IV infusion Q6W
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of pembrolizumab given in combination with either ipilimumab or placebo as first-line treatment in participants with metastatic non-small cell lung cancer (NSCLC). The primary hypothesis of this study is that overall survival (OS) and/or progression-free survival (PFS) is prolonged in participants who receive pembrolizumab and ipilimumab compared to those who receive pembrolizumab and placebo.

With Amendment 6 (effective date: 11-Dec-2020), active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded. Participants will discontinue ipilimumab and placebo and participants who remain on treatment will receive open-label pembrolizumab only.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of Stage IV metastatic non-small cell lung cancer (NSCLC) (American Joint Committee on Cancer version 8)
* Has measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as determined by investigator
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has a life expectancy of at least 3 months
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Female participants of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female participants of reproductive potential must agree to use contraception starting from the first dose of study medication, throughout the study period, and for up to 120 days after the last dose of study medication

Exclusion Criteria:

* Has received prior systemic chemotherapy/other targeted or biological antineoplastic therapy treatment for their Stage IV metastatic NSCLC
* Has a tumor that harbors an epidermal growth factor receptor (EGFR)-sensitizing (activating) mutation or an anaplastic lymphoma kinase (ALK) translocation
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study therapy
* Has received prior therapy with an anti-Programmed Cell Death Receptor 1 (PD-1), anti-Programmed Cell Death Receptor Ligand 1 (anti-PD-L1), or anti- Programmed Cell Death Receptor Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior radiotherapy within 2 weeks of start of study therapy or received lung radiation therapy of >30 Gray (Gy) within 6 months of the first dose of study therapy
* Has recovered from all radiation-related toxicities, does not require corticosteroids, and has not had radiation pneumonitis
* Is receiving systemic steroid therapy ≤7 days prior to the first dose of study therapy or receiving any other form of immunosuppressive medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cancers
* Has known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (i.e., doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study therapy
* Has a history of (non-infectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease
* Has had an allogeneic tissue/solid organ transplant
* Has received a live vaccine within 30 days prior to the first dose of study therapy
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B or known active hepatitis C virus infection
* Has a known history of active tuberculosis
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial
* Is a regular user of any illicit drugs or had a recent history of substance abuse
* Is pregnant or breast feeding or expecting to conceive starting from the first dose of study medication, throughout the study period, and for up to 120 days after the last dose of study medication
* Has severe hypersensitivity to pembrolizumab and/or any of its excipients and/or to ipilimumab and/or any of its excipients
* Has a c-ros oncogene 1 (ROS1) mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (187):
- United States (25):
  - Mayo Clinic Cancer Center ( Site 0007), Phoenix, Arizona
  - Disney Family Cancer Center ( Site 0035), Burbank, California
  - Pacific Cancer Care ( Site 0001), Monterey, California
  - John Wayne Cancer Institute ( Site 0021), Santa Monica, California
  - Florida Hospital Cancer Institute ( Site 0009), Orlando, Florida
  - Mercy Health-Paducah Medical Oncology and Hematology ( Site 0018), Paducah, Kentucky
  - New England Cancer Specialists ( Site 0019), Scarborough, Maine
  - Boston Medical Center ( Site 0025), Boston, Massachusetts
  - Lahey Hospital & Medical Center ( Site 0020), Burlington, Massachusetts
  - Holy Name Medical Center ( Site 0022), Teaneck, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 0034), New York, New York
  - The Ohio State University Wexner Medical Center ( Site 0016), Columbus, Ohio
  - Mid Ohio Oncology/Hematology Inc. ( Site 0003), Columbus, Ohio
  - Providence Cancer Institute, Franz Clinic - Eastside ( Site 0031), Portland, Oregon
  - Greenville Health System ( Site 8010), Greenville, South Carolina
  - University of Tennessee Erlanger Oncology & Hematology ( Site 0026), Chattanooga, Tennessee
  - Tennessee Cancer Specialists ( Site 0017), Knoxville, Tennessee
  - Texas Oncology-Arlington South ( Site 8006), Arlington, Texas
  - Texas Oncology-Methodist Dallas Cancer Center ( Site 8000), Dallas, Texas
  - Texas Oncology-Flower Mound ( Site 8007), Flower Mound, Texas
  - Texas Oncology-Longview Cancer Center ( Site 8009), Longview, Texas
  - Northwest Cancer Specialists, P.C. ( Site 8001), Vancouver, Washington
  - Virginia Mason Memorial- North Star Lodge Cancer Center ( Site 0033), Yakima, Washington
  - University of Wisconsin Carbone Cancer Center ( Site 0004), Madison, Wisconsin
  - Medical College of Wisconsin Clinical Cancer Center ( Site 0027), Milwaukee, Wisconsin
- Argentina (8):
  - Centro de Investigaciones Clinicas - Clinica Viedma ( Site 0202), Viedma, Río Negro Province
  - Sanatorio Parque ( Site 0201), Rosario, Santa Fe Province
  - Hospital Aleman ( Site 0208), Buenos Aires
  - Hospital Privado Centro Medico Cordoba ( Site 0206), Córdoba
  - Centro Oncologico Riojano Integral ( Site 0203), La Rioja
  - Sanatorio Britanico ( Site 0205), Rosario
  - Instituto de Oncologia de Rosario ( Site 0200), Rosario
  - Centro Medico San Roque ( Site 0207), San Miguel de Tucumán
- Australia (5):
  - Mater Cancer Care Centre ( Site 2102), South Brisbane, Queensland
  - Fiona Stanley Hospital ( Site 2105), Perth, Western Australia
  - Chris OBrien Lifehouse ( Site 2100), Camperdown
  - The Townsville Hospital ( Site 2103), Douglas
  - St Vincents Hospital Melbourne ( Site 2101), Fitzroy
- Brazil (9):
  - Inst de Medicina Integral Professor Fernando Figueira- IMIP ( Site 0302), Recife, Pernambuco
  - Hospital Nossa Senhora da Conceicao ( Site 0306), Porto Alegre, Rio Grande do Sul
  - Clinica de Hematologia e Oncologia Viver Ltda ( Site 0305), Santa Maria, Rio Grande do Sul
  - Instituto do Cancer de Sao Paulo - ICESP ( Site 0300), São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz ( Site 0311), São Paulo, São Paulo
  - Escola Paulista de Medicina - UNIFESP ( Site 0304), São Paulo, São Paulo
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 0312), Barretos
  - CEPON Centro de Pesquisa Oncológicas ( Site 0307), Florianópolis
  - Hospital do Servidor Publico do Estado ( Site 0308), São Paulo
- Canada (7):
  - Tom Baker Cancer Centre ( Site 0119), Calgary, Alberta
  - CancerCare Manitoba ( Site 0106), Winnipeg, Manitoba
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0115), Chicoutimi, Quebec
  - CISSS de la Monteregie-Centre ( Site 0100), Greenfield Park, Quebec
  - CISSS-CA Hotel-Dieu de Levis ( Site 0108), Lévis, Quebec
  - CIUSSS Ouest de l'Ile - St-Mary's Hospital ( Site 0107), Montreal, Quebec
  - St-Jerome Medical Research Inc ( Site 0113), Saint-Jérôme, Quebec
- Chile (5):
  - Clinica Universidad Catolica del Maule ( Site 0413), Talca, El Maule
  - Soc. Prosalud Montes y Orlandi Ltda (Orlandi Oncologia) ( Site 0401), Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0404), Santiago
  - Instituto Nacional del Cancer ( Site 0406), Santiago
  - Hospital Clinico Vina del Mar ( Site 0400), Viña del Mar
- Colombia (5):
  - Hospital Pablo Tobon Uribe ( Site 0505), Medellín, Antioquia
  - Centro de Investigacion Clinica del Country ( Site 0500), Bogotá
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 0506), Bogotá
  - Oncomedica S.A. ( Site 0502), Montería
  - Instituto Cancerologico de Narino Ltda ( Site 0504), Pasto
- France (9):
  - Hopital Nord du Marseille ( Site 0808), Marseille, Cedex 20
  - Institut Bergonie ( Site 0803), Bordeaux
  - CHU de Brest. Hopital Morvan ( Site 0800), Brest
  - Centre Hopitalier Intercommunal Creteil ( Site 0802), Créteil
  - Centre Hospitalier Le Mans ( Site 0804), Le Mans
  - C.H.R.U de Lille - Hopital Calmette ( Site 0805), Lille
  - Hopital Tenon ( Site 0810), Paris
  - Nouvel Hopital Civil ( Site 0809), Strasbourg
  - CHU de Toulouse - Hopital Larrey ( Site 0801), Toulouse
- Germany (8):
  - Evangelische Lungenklinik Berlin ( Site 0903), Berlin
  - Vivantes Klinikum Spandau ( Site 0910), Berlin
  - HELIOS Klinikum Emil von Behring ( Site 0905), Berlin
  - SRH Waldklinikum Gera GmbH ( Site 0907), Gera
  - LungenClinic Grosshansdorf GmbH ( Site 0908), Großhansdorf
  - Universitaetsklinikum Heidelberg ( Site 0900), Heidelberg
  - Universitaetsklinikum Leipzig ( Site 0919), Leipzig
  - Universitaetsklinikum Schleswig Holstein. ( Site 0918), Lübeck
- Hungary (9):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 1502), Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 1506), Budapest
  - Orszagos Onkologiai Intezet ( Site 1509), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 1511), Debrecen
  - Veszprem Megyei Tudogyogyintezet ( Site 1503), Farkasgyepű
  - Petz Aladar Megyei Oktato Korhaz ( Site 1505), Győr
  - Bekes Megyei Pandy Kalman Korhaz. ( Site 1507), Gyula
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz ( Site 1504), Székesfehérvár
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 1501), Szolnok
- Ireland (3):
  - Beaumont Hospital ( Site 1312), Dublin
  - St James Hospital ( Site 1401), Dublin
  - University Hospital Limerick ( Site 1403), Limerick
- Italy (8):
  - IRCCS Casa Sollievo della Sofferenza ( Site 1009), San Giovanni Rotondo (FG), Foggia
  - Humanitas Research Hospital ( Site 1004), Rozzano, Milano
  - Ospedale Mater Salutis ( Site 1005), Legnago, Verona
  - ASST Spedali Civili ( Site 1001), Brescia
  - Istituto Europeo di Oncologia ( Site 1007), Milan
  - Ospedale San Gerardo ASST Monza ( Site 1002), Monza
  - AORN dei Colli Plesso Monaldi ( Site 1003), Napoli
  - Ospedale Santa Maria della Misericordia ( Site 1008), Perugia
- Latvia (2):
  - Pauls Stradins Clinical University Hospital ( Site 1100), Riga
  - Riga East Clinical University Hospital ( Site 1111), Riga
- Mexico (6):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0603), Guadalajara, Jalisco
  - Avix Investigacion Clinica S.C. ( Site 0600), Monterrey, N.L.
  - Medical Care and Research S.A. de C.V. ( Site 0602), Mérida, Yucatán
  - Grupo Medico Camino SC ( Site 0607), Mexico City
  - Medica Sur S.A.B de C.V. ( Site 0608), Mexico City
  - Oncologica de Puebla SA de CV ( Site 0606), Puebla City
- Peru (6):
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 0705), La Victoria, Lima region
  - Centro Especializado de Enfermedades Neoplasicas SRL-CEEN SRL ( Site 0710), Arequipa
  - Instituto Regional de Enfermedades Neoplasicas del Sur IRENSUR ( Site 0704), Arequipa
  - Clinica Internacional Sede San Borja ( Site 0701), Lima
  - Hospital Nacional Cayetano Heredia ( Site 0706), Lima
  - Clinica Peruano Americana S.A. ( Site 0703), Trujillo
- Poland (8):
  - Dolnoslaskie Centrum Onkologii. ( Site 1616), Wroclaw, Lower Silesian Voivodeship
  - Szpital Wojewodzki w Koszalinie im. Mikolaja Kopernika ( Site 1614), Koszalin, West Pomeranian Voivodeship
  - Powiatowe Centrum Zdrowia w Brzezinach ( Site 1615), Brzeziny
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 1609), Bydgoszcz
  - Przychodnia Lekarska Komed ( Site 1602), Konin
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc ( Site 1607), Olsztyn
  - MED-POLONIA Sp. z o.o. ( Site 1605), Poznan
  - Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie ( Site 1600), Warsaw
- South Africa (9):
  - Universitas Annex National Hospital ( Site 1800), Bloemfontein, Free State
  - Clinton Onclogy Clinic ( Site 1804), Alberton, Gauteng
  - Wilgers Oncology Centre ( Site 1808), Pretoria, Gauteng
  - Vincent Pallotti Hospital ( Site 1811), Cape Town
  - University of Stellenbosch and Tygerberg Hospital ( Site 1810), Cape Town
  - Dr G.A. Landers Specialist Oncologist ( Site 1803), Durban
  - Charlotte Maxeke Johannesburg Academic Hospital ( Site 1806), Johannesburg
  - Sandton Oncology Medical Group PTY LTD ( Site 1807), Johannesburg
  - GVI Oncology Clinical Research Centre ( Site 1802), Kraaifontein
- South Korea (4):
  - Seoul National University Hospital ( Site 2303), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2300), Seoul
  - Asan Medical Center ( Site 2302), Seoul
  - Samsung Medical Center ( Site 2301), Seoul
- Spain (7):
  - Hospital Germans Trias i Pujol ( Site 1207), Badalona, Barcelona
  - Hospital Duran i Reynals ( Site 1201), L'Hospitalet de Llobregat, Barcelona
  - Hospital San Pedro de Alcantara ( Site 1208), Cáceres, Extremadura
  - Hospital Universitario Insular de Gran Canaria ( Site 1203), Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitari Vall d Hebron ( Site 1211), Barcelona
  - Hospital Fundacion Jimenez Diaz - Clin. Concepcion ( Site 1209), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1200), Seville
- Taiwan (7):
  - Changhua Christian Hospital ( Site 2406), Changhua
  - Chang Gung Medical Foundation - Kaohsiung ( Site 2404), Kaohsiung City
  - China Medical University Hospital ( Site 2403), Taichung
  - National Cheng Kung University Hospital ( Site 2401), Tainan
  - National Taiwan University Hospital ( Site 2400), Taipei
  - Mackay Memorial Hospital ( Site 2405), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 2402), Taoyuan District
- Thailand (6):
  - Ramathibodi Hospital. ( Site 2563), Ratchthevee, Bangkok
  - Bangkok Hospital Chiangmai ( Site 2560), Mueang, Chiang Mai
  - Chulalongkorn Hospital ( Site 2561), Bangkok
  - Pramongkutklao Hospital ( Site 2564), Bangkok
  - Siriraj Hospital ( Site 2562), Bangkok
  - Khon Kaen University ( Site 2565), Khon Kaen
- Turkey (Türkiye) (12):
  - Acibadem Adana Hastanesi ( Site 1904), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1908), Ankara
  - Uludag Universitesi Tip Fakultesi ( Site 1914), Bursa
  - Ankara Sehir Hastanesi ( Site 1903), Cankaya - Ankara
  - Trakya Uni. Tip Fakultesi ( Site 1911), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1906), Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 1912), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 1901), Izmir
  - Medical Park Izmir Hospital ( Site 1900), Izmir
  - Kocaeli Universitesi Tip Fakultesi ( Site 1909), Kocaeli
  - Inonu Universitesi Tip Fakultesi ( Site 1907), Malatya
  - Karadeniz Teknik Universitesi ( Site 1910), Trabzon
- Ukraine (10):
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council ( Site 2005), Kryviy Rih, Dnipropetrovsk Oblast
  - Cherkasy Regional Hospital ( Site 2020), Cherkasy
  - Regional Clinical Onco Dispensary_ State Medical University ( Site 2012), Chernivtsy
  - Dnipropetrovsk City Multidiscipline Clinical Hosp.4 of DRC ( Site 2000), Dnipropetrovsk
  - MI Prykarpatskyi Clinical Oncology Centrum ( Site 2009), Ivano-Frankivsk
  - PP PPC Acinus Medical and Diagnostic Centre ( Site 2002), Kropyvnytskyi
  - National Cancer Institute of the MoH of Ukraine ( Site 2015), Kyiv
  - Kyiv City Clinical Oncological Center ( Site 2014), Kyiv
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 2003), Lviv
  - MI Odessa Regional Oncological Centre ( Site 2004), Odesa
- United Kingdom (9):
  - Royal Cornwall Hospital ( Site 1325), Truro, Cornwall
  - The Royal Marsden NHS Foundation Trust. ( Site 1326), Sutton, Surrey
  - Belfast City Hospital ( Site 1302), Belfast
  - Royal Free NHS Foundation Trust ( Site 1324), London
  - St. Georges University Hospital NHS Foundation Trust ( Site 1321), London
  - The Royal Marsden NHS Foundation Trust.. ( Site 1327), London
  - The Christie NHS Foundation Trust ( Site 1301), Manchester
  - Mount Vernon Cancer Centre ( Site 1307), Northwood
  - Royal Wolverhampton Hospitals NHS Trust ( Site 1323), Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pd
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Boyer M, Sendur MAN, Rodriguez-Abreu D, Park K, Lee DH, Cicin I, Yumuk PF, Orlandi FJ, Leal TA, Molinier O, Soparattanapaisarn N, Langleben A, Califano R, Medgyasszay B, Hsia TC, Otterson GA, Xu L, Piperdi B, Samkari A, Reck M; KEYNOTE-598 Investigators. Pembrolizumab Plus Ipilimumab or Placebo for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50%: Randomized, Double-Blind Phase III KEYNOTE-598 Study. J Clin Oncol. 2021 Jul 20;39(21):2327-2338. doi: 10.1200/JCO.20.03579. Epub 2021 Jan 29. PMID 33513313
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 568 participants randomized to the study, 563 received at least one dose of study treatment (All Treated Population) and were evaluable for all safety analysis.
Groups:
- Pembrolizumab + Ipilimumab: Participants received 200 mg of pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus 1 mg/kg of ipilimumab by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment. Per Amendment (AM) 6, (effective date: 11-Dec-2020), participants discontinued ipilimumab and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
- Pembrolizumab + Placebo: Participants received 200 mg of pembrolizumab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus placebo by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment. Per Amendment (AM) 6, (effective date: 11-Dec-2020), participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
Period: Overall Study
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Started | 284 | 284
Completed | 0 | 0
Not Completed | 284 | 284
Not completed — Death | 191 | 192
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Sponsor Decision | 90 | 89
Not completed — Laryngeal carcinoma | 0 | 1
Not completed — Not Reported | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 284 | 284 | 568
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.3) | 64.5 (8.8) | 64.1 (9.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 202 | 191 | 393
  Female | 82 | 92 | 174
  Undifferentiated | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 37 | 91
  Not Hispanic or Latino | 208 | 225 | 433
  Unknown or Not Reported | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 33 | 31 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 218 | 223 | 441
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 22 | 22 | 44
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants]
  0 = Fully active; no performance restrictions | 101 | 104 | 205
  1 = Strenuous physical activity restricted; fully ambulatory & able to carry out light work | 183 | 180 | 363
Tumor histology [Count of Participants; unit: Participants]
  Squamous | 77 | 81 | 158
  Non squamous | 207 | 203 | 410
Geographic region [Count of Participants; unit: Participants]
  East Asia | 32 | 31 | 63
  Non-East Asia | 252 | 253 | 505

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of analysis were censored at the date of last known contact. The median survival (in months) and the associated 95% confidence intervals (CIs) were reported using Kaplan-Meier method was used. Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and predominant tumor history (squamous versus non-squamous) was used to estimate hazard ratio (HR) and 95% CIs for first course study treatment per protocol.
Time Frame: Up to approximately 32 months (through data cut-off date: 01 Sep 2020)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 284 | 284
Months | 21.4 [16.6 to NA] — NA = Upper limit OS was not reached at the time of last disease assessment due to insufficient number of participants with events. | 21.9 [18.0 to NA] — NA = Upper limit OS was not reached at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Ipilimumab vs Pembrolizumab + Placebo; Test type: Other; p = 0.74156, Log Rank — One-sided p-value based on log-rank test stratified by ECOG, geographic region of the enrolling site, and predominant tumor history; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.85 to 1.37] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, geographic region of the enrolling site, and predominant tumor history

2. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Based on Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in sum of diameters of target lesions. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The median survival (in months) and associated 95% CIs were reported using Kaplan-Meier method. Cox regression model with Efron's method of tie handling with treatment as covariate stratified by ECOG performance status (0 vs. 1), geographic region of the enrolling site (East Asia vs. non-East Asia), and predominant tumor history (squamous vs. non-squamous) was used to estimate HR and 95% CIs for first course study treatment per protocol.
Time Frame: Up to approximately 32 months (through data cut-off date 01 Sep 2020)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 284 | 284
Months | 8.2 [6.0 to 10.5] | 8.4 [6.3 to 10.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Ipilimumab vs Pembrolizumab + Placebo; Test type: Other; p = 0.71720, Log Rank; One-sided p-value based on log-rank test stratified by ECOG, geographic region of the enrolling site, and predominant tumor history; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.86 to 1.30] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, geographic region of the enrolling site and predominant tumor history

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 Based on BICR
Description: ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by BICR. In this study, RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. Per protocol the ORR was calculated using the Miettinen & Nurminen method stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and predominant tumor history (squamous versus non-squamous) for the first course of study treatment.
Time Frame: Up to approximately 32 months (data cut-off date 01 Sep 2020)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 284 | 284
Percentage of Participants | 45.4 [39.5 to 51.4] | 45.4 [39.5 to 51.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Ipilimumab vs Pembrolizumab + Placebo; Test type: Other; p = 0.50644, Miettinen & Nurminen method; One-sided p-value for testing; Difference in percentage = -0.1, 95% CI 2-sided [-8.2 to 8.1] — Based on Miettinen & Nurminen method stratified by ECOG, geographic region of the enrolling site and predominant tumor history

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 Based on BICR
Description: For participants who demonstrated a confirmed CR (Disappearance of all target lesions) or confirmed PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data. Per protocol, the DOR for all participants who experienced a CR or PR was presented for the first course of study treatment.
Time Frame: Up to approximately 32 months (data cut-off date 01 Sep 2020)
Population: All randomized participants with confirmed complete response or partial response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 129 | 129
Months | 16.1 [12.7 to 26] | 17.3 [14.8 to NA] — NA = DOR 95%CI upper limit not reached at the time of last disease assessment due to insufficient number of participants with events.

5. Secondary Outcome: Time to True Deterioration (TTD) in Cough, Pain in Chest, and Shortness of Breath
Description: TTD was defined as the time to the first onset of a 10-point or greater score deterioration from baseline in any one of the 3 symptoms (cough, pain in chest or shortness of breath), confirmed by a second adjacent 10-point or greater score deterioration from baseline. Cough was based on EORTC QLQ-LC13 question 1, pain in chest was based on EORTC QLQ-LC13 question 10, and shortness of breath was based on EORTC QLQ-C30 question 8. Per protocol, TTD was reported for first course study treatment.
Time Frame: Up to approximately 32 months (data cut-off date 01 Sep 2020)
Population: All participants randomized who received at least one dose of study treatment and had at least one EORTC QLQ-LC13 and EORTC QLQ-C30 available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 268 | 270
Months | NA [12.9778 to NA] — NA = Median TTD and upper limit for TTD was not reached at the time of last disease assessment due to insufficient number of participants with events. | 20.0416 [12.7149 to NA] — NA = Upper limit for TTD was not reached at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Ipilimumab vs Pembrolizumab + Placebo; Test type: Other; p = 0.9112, Log Rank; Two-sided p-value based on log-rank test stratified by ECOG, geographic region of the enrolling site, and predominant tumor histology; Hazard Ratio (HR) = 0.9815, 95% CI 2-sided [0.7386 to 1.3042] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG, geographic region of the enrolling site, and predominant tumor histology

6. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Per protocol, the number of participants who experienced an AE were reported for the first course of study treatment and follow up.
Time Frame: Up to approximately 27 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 282 | 281
Participants | 272 | 263

7. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Per protocol, the number of participants who discontinued study treatment due to an AE were reported for the first course of study treatment.
Time Frame: Up to approximately 24 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 282 | 281
Participants | 105 | 57

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Scale Score to Week 18
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. Per protocol, the change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score were presented for first course study treatment.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study treatment and had at least one EORTC QLQ-C30 assessment available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Ipilimumab | Pembrolizumab + Placebo
Number analyzed (Participants) | 279 | 280
Score on a scale | 3.72 [0.91 to 6.53] | 4.14 [1.42 to 6.86]
Statistical Analysis 1: Comparison: Pembrolizumab + Ipilimumab vs Pembrolizumab + Placebo; Test type: Other; p = 0.8151, cLDA Model; Constrained longitudinal data analysis (cLDA) Model; Difference in LS Means = -0.42, 95% CI 2-sided [-3.96 to 3.12] — Based on a cLDA model with PRO scores as response variable, with covariates for treatment by time interaction, and stratification factors (ECOG, geographic region of the enrolling site, & predominant tumor histology) as covariates

ADVERSE EVENTS:
Time Frame: Up to approximately 56 months
Description: All-cause mortality was reported on all randomized participants (first and second course). Serious and non-serious AEs were reported among participants who received at least one dose of study treatment. MedDRA preferred terms 'Neoplasm progression', 'Malignant neoplasm progression' and 'Disease progression' not related to the drug were excluded. Pembrolizumab + Ipilimumab (second course) was not reported since no participants were eligible for second course treatment.
Groups:
- Pembrolizumab+Ipilimumab (First Course): Participants received 200 mg of pembrolizumab by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus 1 mg/kg of ipilimumab by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment. Per Amendment (AM) 6, (effective date: 11-Dec-2020), participants discontinued ipilimumab and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
- Pembrolizumab+Placebo (First Course); Pembrolizumab + Placebo (Second Course): Participants received 200 mg of pembrolizumab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles of treatment plus placebo by IV infusion on Day 1 of each 6-week cycle for up to 18 cycles of treatment. Per Amendment (AM) 6, (effective date: 11-Dec-2020), participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only.
Arm/Group | Pembrolizumab+Ipilimumab (First Course) | Pembrolizumab+Placebo (First Course) | Pembrolizumab + Placebo (Second Course)
All-Cause Mortality (participants affected / at risk) | 191/284 | 188/284 | 4/18
Serious Adverse Events (participants affected / at risk) | 146/282 | 114/281 | 4/18
Other Adverse Events (participants affected / at risk) | 251/282 | 232/281 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Ipilimumab (First Course) (N=282) | Pembrolizumab+Placebo (First Course) (N=281) | Pembrolizumab + Placebo (Second Course) (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 5 (5) | 3 (3) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Ophthalmoplegia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 7 (10) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 4 (4) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 2 (3) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis migration (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestatic liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 21 (24) | 20 (24) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Autoimmune encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 10 (10) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Ipilimumab (First Course) (N=282) | Pembrolizumab+Placebo (First Course) (N=281) | Pembrolizumab + Placebo (Second Course) (N=18)
Anaemia (Blood and lymphatic system disorders) | 40 (50) | 40 (57) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (5) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 25 (26) | 18 (26) | 1 (1)
Hypophysitis (Endocrine disorders) | 8 (8) | 2 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 43 (48) | 34 (37) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 39 (46) | 52 (57) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 70 (105) | 46 (74) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 15 (17) | 18 (19) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 51 (67) | 40 (51) | 0 (0)
Vomiting (Gastrointestinal disorders) | 30 (44) | 27 (35) | 0 (0)
Asthenia (General disorders) | 51 (66) | 44 (60) | 0 (0)
Chest pain (General disorders) | 15 (15) | 27 (31) | 1 (1)
Fatigue (General disorders) | 47 (66) | 50 (58) | 1 (1)
Oedema peripheral (General disorders) | 24 (31) | 13 (14) | 0 (0)
Pyrexia (General disorders) | 34 (40) | 27 (34) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Cystitis (Infections and infestations) | 5 (6) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 15 (16) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 16 (17) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (20) | 15 (19) | 0 (0)
Alanine aminotransferase increased (Investigations) | 31 (41) | 20 (26) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 37 (44) | 15 (15) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 20 (22) | 12 (13) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 16 (22) | 16 (22) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (8) | 3 (4) | 1 (2)
Blood phosphorus decreased (Investigations) | 0 (0) | 4 (5) | 1 (1)
C-reactive protein increased (Investigations) | 4 (4) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 9 (9) | 10 (12) | 1 (1)
Weight decreased (Investigations) | 29 (33) | 26 (29) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 61 (73) | 39 (44) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (25) | 16 (25) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (15) | 18 (29) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (9) | 3 (3) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 8 (17) | 7 (14) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (21) | 6 (6) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (30) | 16 (28) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (13) | 11 (14) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (22) | 14 (19) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (7) | 7 (9) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (46) | 45 (55) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (36) | 29 (34) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (22) | 21 (25) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 14 (14) | 18 (20) | 0 (0)
Anxiety (Psychiatric disorders) | 8 (10) | 16 (19) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (23) | 23 (24) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (53) | 58 (77) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (49) | 44 (51) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 24 (27) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 18 (20) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 8 (12) | 7 (8) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15) | 18 (18) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 69 (99) | 58 (78) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 57 (78) | 45 (63) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 24 (29) | 12 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03302234/Prot_SAP_000.pdf